CLINICAL TRIAL: NCT02674932
Title: Assessment of a Character Strengths Intervention in Improving Treatment Outcomes Among Psychiatrically Hospitalized Youth
Brief Title: Character Strengths Intervention Among Psychiatrically Hospitalized Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Paresh Patel, Clinical Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HUM00107976
Record Dates: First submitted 2016-01-29; First posted 2016-02-05 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Psychiatric Hospitalization; Mental Disorders; Child/Adolescent Problems
MeSH Terms: conditions — Mental Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Signature Strengths (Experimental): Patients will complete the Values in Action Youth Survey (VIA-Youth) and will receive a list of his/her top character strengths ("signature strengths"). The patient will then participate in the Identifying and Using Signature Strengths Intervention.
  Interventions: Behavioral: Identifying and Using Signature Strengths
- Coping Skills + Memory Aid (Active Comparator): Patients will complete the VIA-Youth but will not receive any results. The patient will then participate in the Identifying and Writing Down Coping Skills Intervention.
  Interventions: Behavioral: Identifying and Writing Down Coping Skills
- Coping Skills (Treatment as Usual) (Other): Patients will complete the VIA-Youth but will not receive any results. After completing the VIA-Youth, the study team member and patient will have a treatment-as-usual discussion about coping skills. (This is equivalent to treatment as usual that is already provided on the psychiatric unit-doctors and nurses on the unit already have this a discussion about coping skills with patients).
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Identifying and Using Signature Strengths — The purpose of the intervention is to identify and focus on one's morally valued strengths and utilize them (i.e. incorporate them into coping skills) to overcome challenges. The study team member and patient will discuss each top strength and ways to use them as coping skills. The patient will identify 2-4 coping mechanisms per strength, and will write his/her strengths and self-identified coping skills on index cards.
  Arms: Signature Strengths
Behavioral: Identifying and Writing Down Coping Skills — The study team member and patient will discuss the importance of having coping skills to deal with stressful and difficult situations. The patient will then identify at least six coping skills and write them down on index cards.
  Arms: Coping Skills + Memory Aid
Behavioral: Treatment as Usual — The study team member and patient will discuss the importance of having coping skills to deal with stressful and difficult situations. The patient will then identify coping skills that could be helpful (but will not write them down).
  Arms: Coping Skills (Treatment as Usual)

SUMMARY:
Research has shown that identifying and using one's character strengths in new ways decreases depressive symptoms and increases happiness in adults in the general population. Recently, we found that a similar intervention increases the self-esteem and self-efficacy of children and adolescents being treated in an inpatient psychiatric unit. The purpose of this study is to better understand the effects that discovering one's character strengths and incorporating them into coping skills will have on treatment outcomes in patients admitted to a child and adolescent inpatient psychiatric unit.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate whether a character strengths-based intervention results in significant improvements in measures of depression, anxiety, resiliency, optimism, self-perception, and life-satisfaction of psychiatrically hospitalized youth up to three months following admission. Secondary aims are to: (1) examine participants' strengths profile to identify potential correlates between character strengths, psychiatric diagnoses and intervention effectiveness; and (2) determine whether patients who continue to incorporate their strengths into coping skills at follow-up assessments exhibit greater improvement over-time.

Participants will be 210 adolescents aged 12 to 17 years admitted to the Child and Adolescent Psychiatric Inpatient Program and will be randomized into one of the three groups. All participants will complete the Values in Action Inventory of Strengths for Youth (VIA-Youth) Survey on their second hospital day and subsequently receive the signature strengths intervention (experimental group), coping skills with memory aids comparison exercise (positive control group), or coping skills without memory aids (treatment-as-usual control group). Outcome measures will be completed by all participants at baseline (day 1 on unit), post-treatment (day 4 on unit), and 1- and 3-months following admission. The proposed research represents a change in paradigm, as we aim to specifically examine the therapeutic benefit of the positive psychology element of our intervention conducted in the pilot study among youth with severe mental illness.

ELIGIBILITY:
Inclusion Criteria:

* Patient on Child and Adolescent Psychiatric Unit

Exclusion Criteria:

* Cognitive disability or severe psychosis preventing understanding of survey measures
* Prior use of VIA-Youth Survey
* Absence of legal guardian to consent

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in depression symptoms over time compared to baseline | baseline, 3 days, 1 month, 3 months
  Depression will be measured using Patient Health Questionnaire (PHQ) for adolescents, and percent change in depression score will be compared across the 3 arms.
Change in anxiety symptoms over time compared to baseline | baseline, 3 days, 1 month, 3 months
  Anxiety will be measured using the 5-item Screen for Child Anxiety Related Emotional Disorders (SCARED), and percent change in anxiety score will be compared across the 3 arms.

SECONDARY OUTCOMES:
Change in self-esteem over time compared to baseline | baseline, 3 days, 1 month, 3 months
  Self-esteem will be measured using the Rosenberg Self-Esteem Scale (SES), and percent change in self-esteem score will be compared across the 3 arms.
Change in self-efficacy over time compared to baseline | baseline, 3 days, 1 month, 3 months
  Self-efficacy will be measured using the General Self-Efficacy Scale (GSE), and percent change in self-efficacy score will be compared across the 3 arms.
Change in resiliency over time compared to baseline | baseline, 3 days, 1 month, 3 months
  Resiliency will be measured using the 10-item Connor Davidson Resiliency Scale (CD-RISC-10), and percent change in resiliency score will be compared across the 3 arms.
Change in life-satisfaction over time compared to baseline | baseline, 3 days, 1 month, 3 months
  Life satisfaction will be measured using the Brief Multidimensional Students' Life Satisfaction Scale - PTPB version (BMSLSS-PTPB), and percent change in life satisfaction score will be compared across the 3 arms.

CONTACTS AND LOCATIONS:
Overall Officials: Paresh D Patel, MD, PhD, Principal Investigator — Department of Psychiatry, University of Michigan

IPD SHARING:
Plan to Share IPD: No